CLINICAL TRIAL: NCT00737659
Title: Phase IV, Open-Label, Multicenter, Randomized Study Comparing Mycophenolate Mofetil (MMF) Dose Adjustment Based on Blood MPA Concentration to Standard Care Treatment With MMF in Renal Transplant Recipients Receiving Tacrolimus
Brief Title: CellCept® Dose Adjustment Versus Fixed Dose (Standard Care) in Renal Transplant Recipients
Acronym: MMF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Eytan Mor Prof., Rabin MC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21706
Record Dates: First submitted 2008-08-17; First posted 2008-08-19 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2008-12

CONDITIONS: Renal Transplant
Keywords: Renal Transplant; Renal; Transplant; MMF; MPA; Recipients
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Concentration Controlled (CC)group will receive an individually adjusted MMF dosing regimen based on the plasma concentrations of mycophenolic acid (MPA,the active metabolite of mycophenolate mofetil).
  Interventions: Drug: Mycophenolate mofetil (CellCept® )
- 2 (Active Comparator): Fixed dose (FD) group will receive an a priori set dose of 2mg\day MMF, the recommended dose, with a possible secondary adaptation by the clinician based on criteria of clinical efficacy, toxicity or interactions with other medications.
  Interventions: Drug: Mycophenolate mofetil (CellCept® )

INTERVENTIONS:
Drug: Mycophenolate mofetil (CellCept® ) — Concentration Control group: MMF dosage will be adjusted (by addition or subtraction of least 250 mg of MMF twice a day) based on MPA levels (MPA AUC target of 40 mg*h\L) measured on Days 7,14,Months 1,3,6 and 12.
  Other Names: CellCept®; MMF
  Arms: 1
Drug: Mycophenolate mofetil (CellCept® ) — Fixed Dose group, MMF dosage will be adjusted based on standard care
  Arms: 2

SUMMARY:
In order to avoid renal transplant rejection, the immune system should be suppressed. After the renal transplant subjects are treated with a combination of two to four different types of immunosuppressive drugs. Theses drugs are very efficient in the prevention of the renal transplant rejection. Still, they can cause side effect.

Research in renal transplant tries to find the best treatment in order to avoid renal rejection on one hand and to reduce as much as possible the undesired adverse and toxicity effects on the other hand.

Therapeutic efficacy and the onset of adverse effects are influenced by levels of mycophenolic acid (MPA, the active metabolite of MMF, CellCept®).

The primary objective of this study is to assess the treatment superiority of CellCept® Dose Adjustment treatment, based on individual MPA concentration value monitored periodically, against treatment with CellCept® Fixed Dose (standard care).

DETAILED DESCRIPTION:
Patient will be randomized into two treatment groups on a 1:1 ratio. Both groups will be treated with the same drugs which is the usual treatment for avoiding renal transplant rejection. In one group the CellCept® dose will be adjusted based on MPA concentration value which will be monitored periodically; and the second group will be treated with CellCept® Fixed Dose (based on the clinical judgment of the treating physician).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, between 18 to 70 years of age at the time of enrollment.
* Patient who received first or second renal transplant.
* Patients who are 0-14 days post transplant.
* Patients capable of understanding the purposes and risks of the study who signed a written informed consent to participate and to comply with the requirements of the study.

Exclusion Criteria:

* Women lactating, pregnant or of childbearing potential not using a reliable contraceptive method before beginning study drug therapy, during therapy and for 4 months following their last dose of the study drug therapy.
* Patients with severe diarrhea or other gastrointestinal disorders that might interfere with their ability to absorb oral medication, including diabetic patients with previously diagnosed diabetic gastroenteropathy.
* Patients with a history of a psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study.
* Patients with evidence of an active systemic infection requiring the continued use of antibiotics or evidence of an HIV infection, or the presence of a chronic active hepatitis B (HBs-Ag positive) or C.
* Current or historic Panel Reactive Antibody (PRA) >50%
* Positive crossmatch (irrespective of method).
* Cold ischemia time of the graft of more than 30 hours.
* Patients who had received an investigational new drug within the last three months at the time of enrollment.
* Multi-organ recipients (e.g. kidney and pancreas) or previous transplant with any organ other than kidney.
* Patients with any known hypersensitivity to MPA, EC-MPS or other components of the formulation (e.g. lactose).
* Patients with thrombocytopenia (< 75,000/mm3), with an absolute neutrophil count of <1,500/mm3, and/or leukocytopenia (< 2,500/mm3), and/or hemoglobin < 6 g/dL at Screening or Baseline.
* Patients with a history of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin.
* Previous exposure to EC-MPS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint Treatment failure defined as a biopsy proven acute rejection, graft loss, death, MMF discontinuation or lost to follow-up. | During the first 12 months following randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Eytan Mor, Prof., Principal Investigator — Rabin Medical Center; Richard Nakache, Prof., Principal Investigator — Sorasky Medical Center
Locations (2):
- Israel (2):
  - Rabin Medical Center, Petach Tikvah
  - Tel Aviv sourasky Medical Center, Tel Aviv